CLINICAL TRIAL: NCT00222092
Title: Effect of Octreotide, Somatostatin, Pentoxyfilline or Placebo in the Prevention and the Course of Post-ERCP Pancreatitis and Study of Molecular Markers in Post-ERCP Pancreatitis
Brief Title: Somatostatin, Octreotide, Pentoxyfilline in the Prevention of Post-ERCP Pancreatitis and Molecular Markers
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Other Study IDs: SIG-2005
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2005-09

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: post-ERCP pancreatitis; prophylaxis; prognosis; natural course; molecular markers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Octreotide, somatostatin and pentoxyfilline commercially available drugs that are used in various clinical situations. They are safe and known for years. Octreotide and somatostatin have been used in many studies for the prophylaxis and treatment of pancreatitis and post-ERCP pancreatitis, while pentoxyfilline has shown effect on patients with alcoholic hepatitis, obstructive vasculitis etc. The aim of the study is to evaluate the efficacy of any of those treatments for the prophylaxis and treatment of post-ERCP pancreatitis. In addition some molecular markers of acute and chronic inflammation will be measured before and after the endoscopic procedures according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing endoscopic retrograde cholangiopancreatography

Exclusion Criteria:

* children, pregnant or breastfeeding women
* patients with coagulation disorders
* inability to access the papilla of Vater due to technical difficulties (previous surgery, malignant obstruction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing endoscopic retrograde cholangiopancreatography
Sampling Method: Non-Probability Sample
Enrollment: 300
Dates: Start 2005-09; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Sigounas, MD, Principal Investigator — University of Ioannina
Locations (1):
- Hepato-Gastroenterology Unit, Medical School of Ioannina - Greece, Ioannina, Greece